CLINICAL TRIAL: NCT03461965
Title: The Use of 3D Printed Models in Mohs Micrographic Surgery
Brief Title: 3D Printed Models in Mohs Micrographic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6617; T32AR007569 (NIH)
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Mohs Micrographic Surgery
Keywords: 3D printing; Patient education

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from University Hospitals Department of Dermatology MMS Clinics at the Cleveland Medical Center, Chagrin Highlands and Westlake Locations. These patients will be randomly assigned to a control (50%) or experimental group (50%) prior to the onset of the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education with 3D printed model (Experimental): The experimental group will be educated on MMS with a standardized script in addition to a 3D MMS model
  Interventions: Behavioral: 3D printed model; Behavioral: Verbal Counselling
- Verbal Counselling (Active Comparator): Participants in the control group will be educated on MMS according to the current standard of care, verbal counselling, with a standardized script
  Interventions: Behavioral: Verbal Counselling

INTERVENTIONS:
Behavioral: 3D printed model — A printed 3D model of MMS will be created showing a model of skin, and a tumor to visually depict the surgery
  Arms: Education with 3D printed model
Behavioral: Verbal Counselling — Participants will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and MMS

SUMMARY:
Patients undergoing Mohs micrographic surgery (MMS) frequently experience anxiety. It has been suggested that enhanced patient education prior to the procedure may decrease patient anxiety. The purpose of the study is to investigate if optimized participant education enhances participant understanding, decreases participant anxiety and increases participant satisfaction.

DETAILED DESCRIPTION:
1. To investigate if participant education with a 3 dimensional printed (3DP) MMS model and standardized script protocol increases participant understanding of MMS more than current standard of care (control group) at the University Hospitals Cleveland Medical Center MMS Clinics.
2. To investigate if participant education with a 3DP MMS model and standardized script protocol decreases perioperative participant anxiety during MMS more than current standard of care (control group) at the University Hospitals Cleveland Medical Center MMS Clinics.
3. To evaluate if participant satisfaction with a 3DP MMS model and standardized script protocol increases participant satisfaction during MMS more than current standard of care (control group) at the University Hospitals Cleveland Medical Center MMS Clinics.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing MMS at University Hospitals Cleveland Medical Center, Chagrin Highlands and Westlake Campus
* Capable of reading and completing all subjective questionnaires

Exclusion Criteria:

* Cannot complete the survey measures independently for any reason

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mann, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Education With 3D Printed Model: The experimental group will be educated on MMS with a standardized script in addition to a 3D MMS model
  3D printed model: A printed 3D model of Mohs Micrographic Surgery will be created showing a model of skin, and a tumor to visually depict the surgery
  Verbal Counselling: patients will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
- Verbal Counselling: Participants in the control group will be educated on MMS according to the current standard of care, verbal counselling, with a standardized script
  Verbal Counselling: patients will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
Period: Overall Study
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Started | 42 | 40
Completed | 42 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Education With 3D Printed Model: The experimental group will be educated on MMS with a standardized script in addition to a 3D MMS model
  3D printed model: A printed 3D model of Mohs Micrographic Surgery will be created showing a model of skin, and a tumor to visually depict the surgery
  Verbal Counselling: patients will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
  Participants in the control group will be educated on MMS according to the current standard of care, verbal counselling, with a standardized script
  Verbal Counselling: patients will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
- Total: Total of all reporting groups
Arm/Group | Education With 3D Printed Model | Verbal Counselling | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.83 (11.34) | 67.83 (12.89) | 67.83 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 24 | 25 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82
Previous MMS experience [Count of Participants; unit: Participants] — Number of patients who previously underwent MMS
  Participants
    Mohs Experience | 20 | 19 | 39
    No Mohs Experience | 22 | 21 | 43
Baseline STAI Y-2 "Trait Anxiety" [Mean (Standard Deviation); unit: units on a scale] — Baseline anxiety from form Y-2 of STAI scale - measures patient's trait or static anxiety
  The STAI is a well-known, frequently used measure of patient anxiety within the clinical setting. This form consists of two forms to assess state anxiety (Y-1) and a participant's baseline trait anxiety (Y-2).
  The Y-2 form consists of 20 Likert-type questions with scores ranging from 20 to 80, with higher scores indicating higher anxiety
  units on a scale | 29.8 (7.53) | 31.1 (8.85) | 30.5 (8.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Correct and Incorrect Mohs Quiz Responses
Description: This is an in-house-designed, short questionnaire with 6 multiple choice objective questions related to the participant's understanding of Mohs. A higher percentage of correct answers indicate a better understanding of Mohs.
  Reported data are percent of responses answered correctly and incorrectly totaled across all participants in each arm
Time Frame: Post surgery (1 day)
Measure: Number; unit: Percent of quiz responses
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Number analyzed (Participants) | 42 | 40
Percent of quiz responses
  Correct Quiz Responses | 93.25 | 85.83
  Incorrect Quiz Responses | 6.75 | 14.17
Statistical Analysis 1: Comparison: Education With 3D Printed Model vs Verbal Counselling; Comparing total responses that were correct across all participants in both arms; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.007, t-test, 2 sided

2. Secondary Outcome: Change in State-Trait Anxiety Inventory (STAI) Y-1 (State Anxiety) Score
Description: The STAI is a well-known, frequently used measure of patient anxiety within the clinical setting. This form consists of two forms to assess state anxiety (Y-1) and a participant's baseline trait anxiety (Y-2).
  The Y-1 form consists of 20 Likert-type questions with scores ranging from 20 to 80, with higher scores indicating higher anxiety. Reported values are change in "state anxiety' (post-stage minus baseline)
Time Frame: From baseline to post surgery (1 day)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Number analyzed (Participants) | 42 | 40
Score on a scale | -4.95 (6.95) | -3.3 (9.37)
Statistical Analysis 1: Comparison: Education With 3D Printed Model; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Verbal Counselling; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p < 0.03, t-test, 2 sided
Statistical Analysis 3: Comparison: Education With 3D Printed Model vs Verbal Counselling; Comparing change in scores (post-stage minus baseline) between experimental and control groups; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.352, t-test, 2 sided; paired t-test

3. Secondary Outcome: Change in Visual Analog Scale (VAS) Anxiety Score
Description: The VAS is a frequently employed Likert-type scale that is used to measure anxiety. This 0-10 scale documents the patients current state of anxiety, with higher scores indicating worse anxietey, and can be answered by patients with an average reading level. Estimated time of completion is under 30 seconds. This form has been used in 2 studies to date and previously by experimental team to assess intraoperative anxiety in Mohs.
Time Frame: From baseline to post surgery (1 day)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Number analyzed (Participants) | 42 | 40
Score on a scale | -1.31 (2.00) | -0.53 (1.54)
Statistical Analysis 1: Comparison: Education With 3D Printed Model; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Verbal Counselling; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.04, t-test, 2 sided
Statistical Analysis 3: Comparison: Education With 3D Printed Model vs Verbal Counselling; Comparing change in scores (post-stage minus baseline) between experimental and control groups; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.052, t-test, 2 sided; paired t-test

4. Secondary Outcome: Change in Visual Analog Scale (VAS) Understanding Score
Description: The VAS is a frequently employed Likert-type scale that because of the ease of use this tool has been converted to assess other objective measures including understanding. This 0-10 scale documents the participant's current state of understanding, with higher scores indicating better understanding, and can be answered by patients with an average reading level. Estimated time of completion is under 30 seconds. This form has been used by experimental team to assess intraoperative understanding in Mohs.
Time Frame: From baseline to post surgery (1 day)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Number analyzed (Participants) | 42 | 40
Score on a scale | 1.83 (2.22) | 2.46 (2.34)
Statistical Analysis 1: Comparison: Education With 3D Printed Model; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Verbal Counselling; Difference of pre (baseline) and post-test scores within each treatment group; Test type: Other — p-value < 0.05 was considered statistically significant; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Education With 3D Printed Model vs Verbal Counselling; Comparing change in scores (post-stage minus baseline) between experimental and control groups; Test type: Other — p-value < 0.05 was considered statistically significant; p = 0.208, t-test, 2 sided; paired t-test

5. Secondary Outcome: Satisfaction Survey Score
Description: Participants were provided 3 subjective questions related to their satisfaction with the explanation of MMS that they received. This scale included questions regarding satisfaction with their explanation of the MMS procedure, if the explanation used could be improved, and if they recommended other patients be provided a similar explanation of MMS, with each question scored from 1 to 5, with higher scores indicating greater satisfaction. Total score range is 0 to 15, with higher scores indicating greater satisfaction.
Time Frame: Post surgery (1 day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education With 3D Printed Model | Verbal Counselling
Number analyzed (Participants) | 42 | 40
score on a scale | 14.69 (0.811) | 13.58 (1.599)
Statistical Analysis 1: Comparison: Education With 3D Printed Model vs Verbal Counselling; Test type: Other — p-value < 0.05 was considered statistically significant; p < 0.03, Chi-squared

ADVERSE EVENTS:
Description: Adverse Events were not collected because no adverse events were expected
Groups:
- Education With 3D Printed Model: The experimental group will be educated on MMS with a standardized script in addition to a 3D MMS model
  3D printed model: A printed 3D model of Mohs Micrographic Surgery will be created showing a model of skin, and a tumor to visually depict the surgery
  Verbal Counselling: Participants will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
- Verbal Counselling: Participants in the control group will be educated on MMS according to the current standard of care, verbal counselling, with a standardized script
  Verbal Counselling: Participants will be educated with a standardized script on skin cancer, risks for skin cancer, treatment options, and Mohs Micrographic Surgery
Arm/Group | Education With 3D Printed Model | Verbal Counselling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03461965/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03461965/ICF_001.pdf